CLINICAL TRIAL: NCT02404415
Title: The Vanderbilt Atrial Fibrillation Ablation Registry
Acronym: VAFAR
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, M. Benjamin Shoemaker, Clinical Instructor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 110881
Record Dates: First submitted 2015-03-19; First posted 2015-03-31 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: catheter ablation; genomics
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Vanderbilt Atrial Fibrillation Ablation registry (VAFAR) is a prospective clinical and genetic biorepository that systematically enrolls patients undergoing atrial fibrillation (AF) ablation. The registry was started in 2011 and has greater than 1000 AF ablation records with stored blood and DNA samples. The goals of VAFAR are to: 1) identify clinical, genetic, and serological predictors of response to AF ablation in order to improve patient selection, and 2) to provide a resource for translational research investigating the electrophysiologic mechanisms of AF pathogenesis.

DETAILED DESCRIPTION:
The study population consists of patients at least 18 years of age who are scheduled for AF ablation at Vanderbilt University. Data recorded at enrollment includes a detailed past medical history and measurements from pre-ablation imaging (cardiac MRI or CT). At the time of ablation, a blood sample is collected for storage of plasma/serum and extraction of DNA, and details of the ablation procedure are recorded. Post-ablation monitoring for arrhythmia recurrence is performed according to a standard clinical follow-up schedule at 3, 6, and 12-months. ECG's are performed at each follow-up visit along with placement of an ambulatory ECG-monitor. At 6-months post-ablation, cardiac imaging with a repeat cardiac MRI or CT is performed.

ELIGIBILITY:
Inclusion criteria:

1. Age >18 years
2. Able to give written, informed consent
3. Scheduled for an ablation procedure to treat atrial fibrillation

Exclusion criteria:

1. None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults scheduled to undergo an atrial fibrillation ablation
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2011-10; Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Moore B Shoemaker, MD, MSCI, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Shoemaker MB, Muhammad R, Farrell M, Parvez B, White BW, Streur M, Stubblefield T, Rytlewski J, Parvathaneni S, Nagarakanti R, Roden DM, Saavedra P, Ellis C, Whalen SP, Darbar D. Relation of morbid obesity and female gender to risk of procedural complications in patients undergoing atrial fibrillation ablation. Am J Cardiol. 2013 Feb 1;111(3):368-73. doi: 10.1016/j.amjcard.2012.10.013. Epub 2012 Nov 17. PMID 23168290
- [Result] Benjamin Shoemaker M, Muhammad R, Parvez B, White BW, Streur M, Song Y, Stubblefield T, Kucera G, Blair M, Rytlewski J, Parvathaneni S, Nagarakanti R, Saavedra P, Ellis CR, Patrick Whalen S, Roden DM, Darbar R D. Common atrial fibrillation risk alleles at 4q25 predict recurrence after catheter-based atrial fibrillation ablation. Heart Rhythm. 2013 Mar;10(3):394-400. doi: 10.1016/j.hrthm.2012.11.012. Epub 2012 Nov 23. PMID 23178686
- [Result] Shoemaker MB, Gidfar S, Pipilas DC, Tamboli RA, Savio Galimberti E, Williams DB, Clements RH, Darbar D. Prevalence and predictors of atrial fibrillation among patients undergoing bariatric surgery. Obes Surg. 2014 Apr;24(4):611-6. doi: 10.1007/s11695-013-1123-8. PMID 24214203
- [Result] Shoemaker MB, Bollmann A, Lubitz SA, Ueberham L, Saini H, Montgomery J, Edwards T, Yoneda Z, Sinner MF, Arya A, Sommer P, Delaney J, Goyal SK, Saavedra P, Kanagasundram A, Whalen SP, Roden DM, Hindricks G, Ellis CR, Ellinor PT, Darbar D, Husser D. Common genetic variants and response to atrial fibrillation ablation. Circ Arrhythm Electrophysiol. 2015 Apr;8(2):296-302. doi: 10.1161/CIRCEP.114.001909. Epub 2015 Feb 14. PMID 25684755
- [Derived] Farrell M, Yoneda Z, Montgomery J, Crawford D, Wray LL, Xu M, Kolek MJ, Richardson T, Lugo R, Metawee M, Michaud G, Estrada JC, Saavedra P, Shen S, Kanagasundram A, Ellis CR, Crossley G, Roden D, Shoemaker MB. Non-pulmonary vein mediated atrial fibrillation: A novel sub-phenotype. PLoS One. 2017 Sep 7;12(9):e0184354. doi: 10.1371/journal.pone.0184354. eCollection 2017. PMID 28880943